CLINICAL TRIAL: NCT00723060
Title: Comparison of Effects Between Conventional Dose and High Dose Escitalopram on Clinical Improvement in Patients With Obsessive-compulsive Disorder (Randomized, Double-blind, Multi-center Study)
Brief Title: Comparison of Effects Between Conventional Dose and High Dose Escitalopram on Clinical Improvement in Patients With Obsessive-compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11769A
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): escitalopram high dose group
  Interventions: Drug: escitalopram
- 2 (Active Comparator): escitalopram conventional group
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — escitalopram high dose group (40mg) escitalopram conventional dose group (20mg)

SUMMARY:
OBJECTIVE: The objective of this study is to compare the effect and safety of conventional dose (20mg) and high dose (40mg) of escitalopram in patients with obsessive-compulsive disorder (OCD).

OVERVIEW OF STUDY DESIGN: Prospective, Randomized, Active-controlled, Double-blind, Multi-center, Clinical Trials STUDY POPULATION: Patients with OCD EFFICACY EVALUATIONS: Y-BOCS (D-YBOCS), HAM-D, HAM-A, CGI-S & -I, GAF, OCI-R SAFETY EVALUATION: Adverse Events / Serious Adverse Events, UKU

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman, aged 18 to 65 years, outpatient
2. Primary OCD patients diagnosed with DSM-IV-TR, having OCD symptoms for more than six months
3. Severity: Y-BOCS score of >= 20 at screening and baseline
4. No history or evidences of clinically significant physical problem, or abnormal laboratory findings at screening
5. Drug free period of at least 2 weeks before study drug administration (in case of fluoxetine, at least 5 weeks). However, allowed medications in this study could be taken even before study drug administration.

Exclusion Criteria:

1. primary active DSM-IV axis I diagnosis other than OCD
2. History of substance, including alcohol, dependence and psychotic symptoms
3. Current depression A. Risk of suicidal attempt B. 20-item Hamilton Depression Rating Scale (HAM-D)(exclude 21th item, obsession) of >17 at screening or baseline
4. Drug allergy A. Known or suspected hypersensitivity to escitalopram or citalopram B. History of severe drug allergic reactions or hypersensitivity
5. History of no response to escitalopram or citalopram treatment
6. History of electroconvulsive therapy or received an injectable antipsychotic formulation within 6 months before screening
7. Women who are pregnant, planning to become pregnant, or breast-feeding
8. Ongoing cognitive behavior therapy (CBT) of OCD
9. Hoarding or collecting type
10. Unable to perform study protocol as clinically assessed by the investigator (ex, severe personality disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The difference of Y-BOCS score average from baseline to 16-week | baseline and16-week

SECONDARY OUTCOMES:
1) CGI-S, CGI-I 2) GAF 3) HAM-D, HAM-A | every 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea